CLINICAL TRIAL: NCT00272961
Title: A Phase 2 Multi-Centre, Randomised, Double-Blind, Placebo Controlled, Dose Ranging Study Of TBC3711 In Subjects With Resistant Hypertension
Brief Title: A Study Of Different Doses Of TBC3711 In Patients With Uncontrolled High Blood Pressure Already Taking Medications For High Blood Pressure.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1341001; GRH01
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-01

CONDITIONS: Resistant Hypertension
MeSH Terms: interventions — N-(2-acetyl-4,6-dimethylphenyl)-3-(3,4-dimethylisoxazol-5-ylsulfamoyl)thiophene-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- ARM 1 (Experimental)
  Interventions: Drug: TBC3711
- ARM 2 (Experimental)
  Interventions: Drug: TBC3711
- ARM 3 (Experimental)
  Interventions: Drug: TBC3711
- ARM 4 (Experimental)
  Interventions: Drug: TBC3711

INTERVENTIONS:
Drug: Placebo — placebo tablet once daily for 12 weeks
  Arms: placebo
Drug: TBC3711 — 10 mg tablets once daily for 10 weeks
  Arms: ARM 1
Drug: TBC3711 — 50 mg tablet once daily for 10 weeks
  Arms: ARM 2
Drug: TBC3711 — 100 mg tablet once daily for 10 weeks
  Arms: ARM 3
Drug: TBC3711 — 200 mg tablet once daily for 10 weeks
  Arms: ARM 4

SUMMARY:
The study was to determine the safe and effective dose of TBC3711 in patients with uncontrolled high blood pressure while already taking blood pressure medications.

DETAILED DESCRIPTION:
The study was stopped due to Pfizer (sponsor) decision that the compound would not be involved in any further clinical development for the indication of resistant hypertension on 05 August 2008. This decision was not based on any safety or efficacy concern.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of resistant hypertension.
* A stable anti-hypertensive drug regimen for at least 30 days.

Exclusion Criteria:

* Sustained blood pressure greater than or equal to 180/120 mmHg.
* Required use of thigh cuff for blood pressure readings.
* Uncontrolled diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Simpsonville, South Carolina
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Carroltown, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1341001&StudyName=A%20study%20of%20different%20doses%20of%20TBC3711%20in%20patients%20with%20uncontolled%20high%20blood%20pressure%20already%20taking%20medications%20for%20high%20blood%20press

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to TBC3711, 4 tablets orally once daily in 2-week placebo run-in phase and 10-week treatment phase.
- TBC3711 10 mg: Participants who received placebo matched to TBC3711 tablet orally once daily in 2-week Placebo Run-in Phase, received TBC3711 10 milligram (mg) tablet and 3 matching placebo tablets orally once daily in 10-week Treatment Phase.
- TBC3711 50 mg: Participants who received placebo matched to TBC3711 tablet orally once daily in 2-week Placebo Run-in Phase, received TBC3711 50 mg tablet and 3 matching placebo tablets orally once daily in 10-week Treatment Phase.
- TBC3711 100 mg: Participants who received placebo matched to TBC3711 tablet orally once daily in 2-week Placebo Run-in Phase, received TBC3711 50 mg tablet and 3 matching placebo tablets orally once daily for 1 week followed by 2 TBC3711 50 mg tablets (equivalent to TBC3711 100 mg) and 2 matching placebo tablets orally once daily for 9 weeks in 10-week Treatment Phase.
- TBC3711 200 mg: Participants who received placebo matched to TBC3711 tablet orally once daily in 2-week Placebo Run-in Phase, received TBC3711 50 mg tablet and 3 matching placebo tablets orally once daily for 1 week followed by 2 TBC3711 50 mg tablets (equivalent to TBC3711 100 mg) and 2 matching placebo tablets orally once daily for 1 week followed by 4 TBC3711 50 mg tablets (equivalent to TBC3711 200 mg) orally once daily for 8 weeks in 10-week Treatment Phase.
Period: Placebo Run-in Phase: Up to Week 2
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Started | 60 | 0 | 0 | 0 | 0
Completed | 49 | 0 | 0 | 0 | 0
Not Completed | 11 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 0 | 0 | 0
Not completed — Subject Defaulted | 5 | 0 | 0 | 0 | 0
Not completed — Participant Needed Prohibited Medication | 2 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 0 | 0 | 0
Period: Treatment Phase: Week 3 Up to Week 12
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Started | 10 | 8 | 11 | 10 | 10
Completed | 8 | 4 | 7 | 7 | 6
Not Completed | 2 | 4 | 4 | 3 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 2
Not completed — Participant Defaulted | 1 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 3 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg | Total
Number analyzed (Participants) | 10 | 8 | 11 | 10 | 10 | 49
Age, Customized [Number; unit: participants]
  18 to 44 Years | 0 | 1 | 0 | 1 | 1 | 3
  45 to 64 Years | 6 | 5 | 10 | 9 | 7 | 37
  Greater Than or Equal to (>=) 65 Years | 4 | 2 | 1 | 0 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5 | 4 | 3 | 17
  Male | 7 | 6 | 6 | 6 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Blood Pressure (BP) Increase
Description: BP is the pressure of the blood within the arteries. It is produced primarily by the contraction of the heart muscle. BP measurement is recorded by 2 numbers: systolic BP (SBP, BP when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle) and diastolic BP (DBP, BP when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles). Maximum increase was calculated by subtracting baseline value from each post-dose measurement and selecting maximum of these values.
Time Frame: Baseline (Pre-Dose on Day 1 of Week 2) up to Week 12
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Here "n" signifies participants evaluable for specified category for each treatment arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Number analyzed (Participants) | 10 | 8 | 11 | 10 | 10
millimeter of mercury (mmHg)
  Sitting SBP (n= 8, 6, 9, 8, 8) | 11.48 (4.04) | 3.10 (4.67) | 11.26 (3.83) | 11.52 (4.03) | 10.46 (4.09)
  Standing SBP (n= 10, 8, 11, 10, 10) | 9.06 (3.24) | 2.96 (3.64) | 8.38 (3.08) | 9.63 (3.23) | 14.76 (3.23)
  Sitting DBP (n= 8, 6, 9, 8, 8) | 8.16 (1.75) | 2.53 (2.02) | 6.73 (1.65) | 1.79 (1.77) | 7.17 (1.81)
  Standing DBP (n= 10, 8, 11, 10, 10) | 7.91 (1.69) | 3.11 (1.90) | 7.11 (1.62) | 2.27 (1.69) | 6.25 (1.74)
Statistical Analysis 1: Comparison: Placebo vs TBC3711 10 mg; Sitting SBP: p-value was obtained using an Analysis of Co-variance (ANCOVA) model on the maximum increase observed with baseline value as a covariate; Test type: Superiority or Other; p = 0.185, ANCOVA; Least Squares (LS) Mean Difference = 8.37, 95% CI 2-sided [-4.21 to 20.96], Standard Error of Mean 6.19
Statistical Analysis 2: Comparison: Placebo vs TBC3711 50 mg; Sitting SBP: p-value was obtained using an ANCOVA model on the maximum increase observed with baseline value as a covariate; Test type: Superiority or Other; p = 0.970, ANCOVA; LS Mean Difference = 0.21, 95% CI 2-sided [-11.16 to 11.59], Standard Error of Mean 5.59
Statistical Analysis 3: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.994, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-11.66 to 11.57], Standard Error of Mean 5.71
Statistical Analysis 4: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.861, ANCOVA; LS Mean Difference = 1.01, 95% CI 2-sided [-10.62 to 12.64], Standard Error of Mean 5.72
Statistical Analysis 5: Comparison: Placebo vs TBC3711 10 mg; Standing SBP: p-value was obtained using an ANCOVA model on the maximum increase observed with baseline value as a covariate; Test type: Superiority or Other; p = 0.221, ANCOVA; LS Mean Difference = 6.10, 95% CI 2-sided [-3.79 to 15.99], Standard Error of Mean 4.90
Statistical Analysis 6: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.880, ANCOVA; LS Mean Difference = 0.68, 95% CI 2-sided [-8.37 to 9.73], Standard Error of Mean 4.49
Statistical Analysis 7: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.900, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-9.78 to 8.63], Standard Error of Mean 4.56
Statistical Analysis 8: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.218, ANCOVA; LS Mean Difference = -5.71, 95% CI 2-sided [-14.91 to 3.50], Standard Error of Mean 4.56
Statistical Analysis 9: Comparison: Placebo vs TBC3711 10 mg; Sitting DBP: p-value was obtained using an ANCOVA model on the maximum increase observed with baseline value as a covariate; Test type: Superiority or Other; p = 0.044, ANCOVA; LS Mean Difference = 5.62, 95% CI 2-sided [0.17 to 11.08], Standard Error of Mean 2.68
Statistical Analysis 10: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.557, ANCOVA; LS Mean Difference = 1.43, 95% CI 2-sided [-3.47 to 6.33], Standard Error of Mean 2.41
Statistical Analysis 11: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.016, ANCOVA; LS Mean Difference = 6.37, 95% CI 2-sided [1.28 to 11.45], Standard Error of Mean 2.50
Statistical Analysis 12: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.695, ANCOVA; LS Mean Difference = 0.99, 95% CI 2-sided [-4.09 to 6.07], Standard Error of Mean 2.50
Statistical Analysis 13: Comparison: Placebo vs TBC3711 10 mg; Standing DBP: p-value was obtained using an ANCOVA model on the maximum increase observed with baseline value as a covariate; Test type: Superiority or Other; p = 0.067, ANCOVA; LS Mean Difference = 4.80, 95% CI 2-sided [-0.36 to 9.95], Standard Error of Mean 2.56
Statistical Analysis 14: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.737, ANCOVA; LS Mean Difference = 0.80, 95% CI 2-sided [-3.96 to 5.55], Standard Error of Mean 2.36
Statistical Analysis 15: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.023, ANCOVA; LS Mean Difference = 5.64, 95% CI 2-sided [0.80 to 10.47], Standard Error of Mean 2.40
Statistical Analysis 16: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.495, ANCOVA; LS Mean Difference = 1.65, 95% CI 2-sided [-3.20 to 6.50], Standard Error of Mean 2.40

2. Primary Outcome: Weighted Mean (Area Under Effect Curve [AUEC]) Blood Pressure Change
Description: AUEC was calculated as the positive area under the change from baseline curve for sitting and standing SBP and DBP to Week 12, estimated by the linear trapezoidal rule corrected for the pre-dose baseline value. In the event that post-dose values returned below baseline at or before Week 12, then AUEC was calculated by setting the negative values to zero and taking only the positive area into account.
Time Frame: Baseline (Pre-Dose on Day 1 of Week 2) up to Week 12
Population: Safety analysis set: all participants who received at least 1 dose of study treatment. "N"(number of participants analyzed): participants evaluable for this measure and n: participants with non-missing baseline and at least 2 non-missing values in treatment phase or in follow-up for specified category for each treatment arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Number analyzed (Participants) | 10 | 7 | 11 | 10 | 10
mmHg
  Sitting SBP (n= 8, 5, 9, 8, 8) | 318.50 (125.20) | 85.91 (158.59) | 214.83 (119.85) | 277.24 (125.27) | 152.10 (126.57)
  Standing SBP (n= 10, 7, 11, 10, 10) | 237.83 (83.52) | 74.79 (99.66) | 122.48 (79.95) | 213.16 (83.46) | 187.24 (83.37)
  Sitting DBP (n= 8, 5, 9, 8, 8) | 256.38 (67.58) | 30.82 (85.41) | 141.61 (63.97) | 31.50 (68.88) | 123.17 (70.03)
  Standing DBP (n= 10, 7, 11, 10, 10) | 282.89 (73.31) | 42.26 (87.57) | 124.90 (70.65) | 27.99 (73.46) | 125.23 (75.08)
Statistical Analysis 1: Comparison: Placebo vs TBC3711 10 mg; Sitting SBP: p-value was obtained using an ANCOVA model on AUEC calculated over treatment and follow-up phases with baseline value as a covariate; Test type: Superiority or Other; p = 0.2577, ANCOVA; LS Mean Difference = 232.59, 95% CI 2-sided [-178.5 to 643.7], Standard Error of Mean 201.83
Statistical Analysis 2: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5552, ANCOVA; LS Mean Difference = 103.67, 95% CI 2-sided [-250.5 to 457.8], Standard Error of Mean 173.86
Statistical Analysis 3: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8174, ANCOVA; LS Mean Difference = 41.26, 95% CI 2-sided [-319.8 to 402.3], Standard Error of Mean 177.26
Statistical Analysis 4: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3557, ANCOVA; LS Mean Difference = 166.40, 95% CI 2-sided [-195.3 to 528.1], Standard Error of Mean 177.55
Statistical Analysis 5: Comparison: Placebo vs TBC3711 10 mg; Standing SBP: p-value was obtained using an ANCOVA model on AUEC calculated over treatment and follow-up phases with baseline value as a covariate; Test type: Superiority or Other; p = 0.2172, ANCOVA; LS Mean Difference = 163.04, 95% CI 2-sided [-99.6 to 425.7], Standard Error of Mean 130.15
Statistical Analysis 6: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.3258, ANCOVA; LS Mean Difference = 115.35, 95% CI 2-sided [-118.8 to 349.5], Standard Error of Mean 116.03
Statistical Analysis 7: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.8352, ANCOVA; LS Mean Difference = 24.67, 95% CI 2-sided [-213.2 to 262.6], Standard Error of Mean 117.88
Statistical Analysis 8: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.6701, ANCOVA; LS Mean Difference = 50.59, 95% CI 2-sided [-187.4 to 288.6], Standard Error of Mean 117.93
Statistical Analysis 9: Comparison: Placebo vs TBC3711 10 mg; Sitting DBP: p-value was obtained using an ANCOVA model on AUEC calculated over treatment and follow-up phases with baseline value as a covariate; Test type: Superiority or Other; p = 0.0466, ANCOVA; LS Mean Difference = 225.57, 95% CI 2-sided [3.6 to 447.5], Standard Error of Mean 108.95
Statistical Analysis 10: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.2274, ANCOVA; LS Mean Difference = 114.77, 95% CI 2-sided [-75.2 to 304.8], Standard Error of Mean 93.2637
Statistical Analysis 11: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.0269, ANCOVA; LS Mean Difference = 224.89, 95% CI 2-sided [27.5 to 422.3], Standard Error of Mean 96.9259
Statistical Analysis 12: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.1780, ANCOVA; LS Mean Difference = 133.22, 95% CI 2-sided [-63.8 to 330.3], Standard Error of Mean 96.7383
Statistical Analysis 13: Comparison: Placebo vs TBC3711 10 mg; Standing DBP: p-value was obtained using an ANCOVA model on AUEC calculated over treatment and follow-up phases with baseline value as a covariate; Test type: Superiority or Other; p = 0.0413, ANCOVA; LS Mean Difference = 240.64, 95% CI 2-sided [9.9 to 471.4], Standard Error of Mean 114.32
Statistical Analysis 14: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.1297, ANCOVA; LS Mean Difference = 157.99, 95% CI 2-sided [-48.3 to 364.3], Standard Error of Mean 102.21
Statistical Analysis 15: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.0185, ANCOVA; LS Mean Difference = 254.90, 95% CI 2-sided [45.0 to 464.8], Standard Error of Mean 104.00
Statistical Analysis 16: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.1382, ANCOVA; LS Mean Difference = 157.66, 95% CI 2-sided [-52.9 to 368.2], Standard Error of Mean 104.33

3. Secondary Outcome: Sitting Systolic Blood Pressure (SBP)
Description: SBP is the BP (pressure exerted by circulating blood on the walls of blood vessels) when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle of heart. A total of 3 measurements were performed and average was calculated at each time point in participant's non-dominant arm using appropriate-sized cuff (cuff bladder encircling at least 80 percent [%] of the arm) after participant sat for 5 minutes for the first measurement and 2 minutes for second and third measurements. The same arm was used throughout the study.
Time Frame: Pre-Dose and 2 hour Post-Dose on Baseline (Day 1 of Placebo Run-In Phase), Week 1, 2, 3, 4, 6, 8, 10
Population: Full analysis set (FAS):all randomized participants who received study treatment at least twice after Placebo Run-in Phase, but not necessarily at 2 consecutive visits. "N" (number of participants analyzed): participants evaluable for this measure, n: participants with non-missing value for specified time-point for each treatment arm, respectively.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Number analyzed (Participants) | 8 | 6 | 9 | 8 | 8
mmHg
  Baseline: Pre-Dose (n= 8, 6, 9, 8, 8) | 158.6 (5.0) | 149.9 (5.6) | 146.5 (4.1) | 151.1 (3.2) | 158.4 (5.8)
  Baseline: Post-Dose (n= 8, 6, 9, 8, 8) | 149.9 (4.9) | 141 (6.4) | 139.7 (6.1) | 149.3 (4.4) | 148.8 (6.4)
  Week 1: Pre-Dose (n= 8, 6, 9, 8, 8) | 156.3 (5.3) | 151 (4.7) | 143.5 (4.9) | 145.3 (4.2) | 154.9 (4.9)
  Week 1: Post-Dose (n= 8, 6, 9, 8, 8) | 151.1 (5.2) | 141.1 (8.8) | 134.4 (5.6) | 139.4 (5.1) | 143.6 (7.4)
  Week 2: Pre-Dose (n= 8, 6, 9, 8, 8) | 149.6 (5.8) | 144.7 (7.5) | 143.5 (5.8) | 147.1 (4.4) | 153.1 (4.5)
  Week 2: Post-Dose (n= 8, 6, 9, 8, 7) | 139.8 (5.5) | 130.6 (10.6) | 134.7 (8.7) | 139 (4.7) | 134.3 (6.9)
  Week 3: Pre-Dose (n= 8, 4, 7, 7, 8) | 148 (4.6) | 141.5 (3.9) | 137.1 (6.5) | 142 (5.2) | 141.8 (6.1)
  Week 3: Post-Dose (n= 8, 5, 6, 7, 8) | 144.2 (4.1) | 138.1 (3.3) | 123.2 (7.5) | 138.5 (6.0) | 130.3 (7.2)
  Week 4: Pre-Dose (n= 7, 5, 8, 8, 8) | 141.4 (4.9) | 141.2 (6.9) | 140.9 (6.9) | 135.8 (3.7) | 140.8 (6.3)
  Week 4: Post-Dose (n= 7, 4, 8, 7, 8) | 143 (5.4) | 137 (4.8) | 132.2 (9.1) | 132.3 (5.1) | 132.8 (10)
  Week 6: Pre-Dose (n= 7, 5, 7, 7, 6) | 149.2 (7.0) | 140.9 (6.2) | 131.7 (4.3) | 137.9 (7.8) | 137.9 (4.6)
  Week 6: Post-Dose (n= 7, 5, 7, 7, 6) | 141.7 (7.4) | 130.9 (3.6) | 124.4 (4.0) | 132.7 (5.7) | 135.3 (8.4)
  Week 8: Pre-Dose (n= 7, 5, 7, 7, 6) | 139.6 (4.7) | 143.2 (6.0) | 126.4 (4.4) | 141.7 (6.9) | 138.3 (5.8)
  Week 8: Post-Dose (n= 7, 5, 7, 7, 6) | 132.7 (6.5) | 136.8 (3.3) | 122.8 (3.4) | 136.6 (5.2) | 125.9 (9.9)
  Week 10: Pre-Dose (n= 7, 4, 7, 7, 6) | 142.1 (6.2) | 148.3 (8.5) | 134.5 (3.2) | 136.8 (5.8) | 141.6 (6.8)
  Week 10: Post-Dose (n= 7, 4, 7, 7, 6) | 134.1 (7.9) | 142 (6.0) | 131.3 (4.1) | 131.7 (6.8) | 132.8 (7.5)

4. Secondary Outcome: Standing Systolic Blood Pressure (SBP)
Description: SBP is the BP (pressure exerted by circulating blood on the walls of blood vessels) when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle of heart. A total of 3 measurements were performed and average was calculated at each time point in participant's non-dominant arm using appropriate-sized cuff (cuff bladder encircling at least 80% of the arm) after participant stood for 2 minutes. The same arm was used throughout the study.
Time Frame: Pre-Dose and 2 hour Post-Dose on Baseline (Day 1 of Placebo Run-In Phase), Week 1, 2, 3, 4, 6, 8, 10
Population: FAS: all randomized participants who received study treatment at least twice after Placebo Run-in Phase, but not necessarily at 2 consecutive visits. Here "N" (number of participants analyzed): participants evaluable for this measure, n: participants with non-missing value for specified time-point for each treatment arm, respectively.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Number analyzed (Participants) | 10 | 8 | 11 | 10 | 10
mmHg
  Baseline: Pre-Dose (n= 10, 8, 11, 10, 10) | 153.6 (4.5) | 147.7 (4.4) | 147.3 (3.3) | 153.8 (4.2) | 154.1 (4.8)
  Baseline: Post-Dose (n= 10, 8, 11, 10, 10) | 146.3 (4.4) | 141.9 (5.5) | 142.4 (4.4) | 149.5 (4.7) | 147 (5.8)
  Week 1: Pre-Dose (n= 10, 8, 11, 10, 10) | 151.5 (5.1) | 147.3 (4.4) | 145.7 (4.3) | 146.8 (4.6) | 154.3 (4.1)
  Week 1: Post-Dose (n= 10, 8, 11, 10, 10) | 147.8 (4.7) | 139.4 (6.9) | 139.2 (5.7) | 141.4 (5.1) | 144.8 (6.8)
  Week 2: Pre-Dose (n= 10, 8, 11, 10, 9) | 151.1 (5.3) | 142.8 (6.3) | 145.8 (4.6) | 150.7 (4.6) | 149.7 (5.1)
  Week 2: Post-Dose (n= 10, 8, 11, 10, 9) | 140.6 (4.8) | 130.8 (7.9) | 138.3 (7.3) | 142.9 (5.1) | 135.8 (6.6)
  Week 3: Pre-Dose (n= 10, 6, 8, 8, 10) | 146.8 (4.1) | 140.9 (2.6) | 136.8 (5.8) | 147.3 (7.1) | 141.2 (6.2)
  Week 3: Post-Dose (n= 10, 7, 7, 8, 10) | 142.4 (3.6) | 137.2 (2.8) | 124.9 (6.4) | 143.1 (7.6) | 128.6 (7.8)
  Week 4: Pre-Dose (n= 9, 7, 9, 9, 10) | 141.8 (4.3) | 139.6 (4.3) | 141.5 (5.8) | 137.4 (5.7) | 139.5 (6.1)
  Week 4: Post-Dose (n= 9, 6, 9, 8, 10) | 141 (4.8) | 133.4 (4.7) | 132.6 (7.7) | 132.6 (5.1) | 129.5 (9.3)
  Week 6: Pre-Dose (n= 9, 7, 8, 8, 8) | 145.3 (5.3) | 138.2 (5.1) | 131.3 (3.5) | 138.9 (8.2) | 134.1 (4.4)
  Week 6: Post-Dose (n= 9, 7, 8, 8, 8) | 139.2 (6.7) | 130.5 (4.4) | 122.8 (4.7) | 130.6 (5.1) | 127.9 (7.2)
  Week 8: Pre-Dose (n= 8, 6, 8, 8, 7) | 139.2 (5.0) | 143.2 (3.2) | 125.9 (4.0) | 141.5 (6.0) | 135.5 (6.1)
  Week 8: Post-Dose (n= 8, 6, 8, 8, 7) | 131.3 (6.6) | 138.6 (2.3) | 124.1 (3.5) | 139.3 (7.4) | 123.3 (9.2)
  Week 10: Pre-Dose (n= 8, 4, 7, 7, 6) | 141.1 (4.6) | 147 (7.4) | 133.4 (3.7) | 137.6 (6.7) | 141 (7.7)
  Week 10: Post-Dose (n= 8, 4, 7, 7, 6) | 133.5 (7.3) | 141.2 (6.3) | 131 (5.3) | 133.5 (8.9) | 128.9 (8.0)

5. Secondary Outcome: Sitting Diastolic Blood Pressure (DBP)
Description: DBP is the BP (pressure exerted by circulating blood on the walls of blood vessels) when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles of heart. A total of 3 measurements were performed and average was calculated at each time point in participant's non-dominant arm using appropriate-sized cuff (cuff bladder encircling at least 80% of the arm) after participant sat for 5 minutes for the first measurement and 2 minutes for second and third measurements. The same arm was used throughout the study.
Time Frame: Pre-Dose and 2 hour Post-Dose on Baseline (Day 1 of Placebo Run-In Phase), Week 1, 2, 3, 4, 6, 8, 10
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Number analyzed (Participants) | 8 | 6 | 9 | 8 | 8
mmHg
  Baseline: Pre-Dose (n= 8, 6, 9, 8, 8) | 95.1 (6.2) | 87 (1.8) | 87.3 (3.0) | 87.8 (3.5) | 99.3 (2.1)
  Baseline: Post-Dose (n= 8, 6, 9, 8, 8) | 91.7 (5.5) | 81 (3.1) | 82.4 (3.8) | 82.7 (3.8) | 93.7 (3.6)
  Week 1: Pre-Dose (n= 8, 6, 9, 8, 8) | 92.6 (5.6) | 88.4 (3.1) | 87.5 (2.8) | 83.6 (4.2) | 99.3 (2.1)
  Week 1: Post-Dose (n= 8, 6, 9, 8, 8) | 89.3 (5.2) | 80.3 (4.0) | 80 (3.5) | 77.6 (4.8) | 94.4 (3.8)
  Week 2: Pre-Dose (n= 8, 6, 9, 8, 8) | 90.6 (5.8) | 86.1 (4.4) | 87.1 (4.0) | 84.4 (4.8) | 96.3 (2.5)
  Week 2: Post-Dose (n= 8, 6, 9, 8, 7) | 83.7 (6.5) | 77.8 (6.5) | 76.3 (5.2) | 71.8 (3.4) | 83.7 (4.8)
  Week 3: Pre-Dose (n= 8, 4, 7, 7, 8) | 89.3 (5.4) | 82.5 (4.4) | 86 (6.7) | 79.8 (7.1) | 91.6 (1.9)
  Week 3: Post-Dose (n= 8, 5, 6, 7, 8) | 87.5 (4.8) | 74.9 (4.1) | 72.8 (4.2) | 71.8 (6.1) | 79.9 (3.2)
  Week 4: Pre-Dose (n= 7, 5, 8, 8, 8) | 83.6 (3.7) | 79.2 (3.8) | 86 (5.3) | 78.1 (4.8) | 89.3 (3.6)
  Week 4: Post-Dose (n= 7, 4, 8, 7, 8) | 82 (3.7) | 74.3 (4.9) | 76.6 (5.7) | 68.6 (3.7) | 81 (4.5)
  Week 6: Pre-Dose (n= 7, 5, 7, 7, 6) | 86.8 (5.3) | 78.9 (3.5) | 78.3 (3.4) | 80.7 (5.2) | 92.1 (3.1)
  Week 6: Post-Dose (n= 7, 5, 7, 7, 6) | 84.1 (5.4) | 73.2 (2.8) | 74.2 (4.2) | 68.9 (3.5) | 84.7 (5.3)
  Week 8: Pre-Dose (n= 7, 5, 7, 7, 6) | 84.8 (5.9) | 82.9 (3.8) | 79.3 (2.7) | 80.6 (5.7) | 93.7 (3.9)
  Week 8: Post-Dose (n= 7, 5, 7, 7, 6) | 78.8 (5.9) | 76.1 (2.6) | 73.2 (3.8) | 73.7 (5.5) | 83.8 (6.1)
  Week 10: Pre-Dose (n= 7, 4, 7, 7, 6) | 87.6 (4.1) | 85.5 (2.2) | 84.8 (3.4) | 79.1 (5.1) | 93 (3.2)
  Week 10: Post-Dose (n= 7, 4, 7, 7, 6) | 79.9 (5.6) | 76.2 (0.9) | 81.3 (3.1) | 66.8 (3.6) | 85.4 (4.4)

6. Secondary Outcome: Standing Diastolic Blood Pressure (DBP)
Description: DBP is the BP (pressure exerted by circulating blood on the walls of blood vessels) when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles of heart. A total of 3 measurements were performed and average was calculated at each time point in participant's non-dominant arm using appropriate-sized cuff (cuff bladder encircling at least 80% of the arm) after participant stood for 2 minutes. The same arm was used throughout the study.
Time Frame: Pre-Dose and 2 hour Post-Dose on Baseline (Day 1 of Placebo Run-In Phase), Week 1, 2, 3, 4, 6, 8, 10
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Number analyzed (Participants) | 10 | 8 | 11 | 10 | 10
mmHg
  Baseline: Pre-Dose (n= 10, 8, 11, 10, 10) | 95.9 (5.1) | 89 (2.7) | 87.9 (2.5) | 90.3 (2.9) | 97.7 (2.8)
  Baseline: Post-Dose (n= 10, 8, 11, 10, 10) | 92.3 (4.8) | 85 (3.3) | 83.1 (3.2) | 85.1 (3.3) | 95.5 (2.9)
  Week 1: Pre-Dose (n= 10, 8, 11, 10, 10) | 95.1 (5) | 90.3 (3.0) | 88.7 (3.0) | 87.2 (4.0) | 98.9 (1.9)
  Week 1: Post-Dose (n= 10, 8, 11, 10, 10) | 91.5 (4.5) | 81.3 (4.7) | 82.7 (3.4) | 81.4 (4.6) | 93.7 (3.1)
  Week 2: Pre-Dose (n= 10, 8, 11, 10, 10) | 92.7 (4.8) | 87.7 (3.8) | 87.9 (3.4) | 89.5 (3.7) | 96.9 (2.6)
  Week 2: Post-Dose (n= 10, 8, 11, 10, 9) | 87.3 (4.8) | 81.4 (5.7) | 80.8 (4.5) | 77.1 (3.2) | 84.8 (4.3)
  Week 3: Pre-Dose (n= 10, 6, 8, 8, 10) | 91.9 (5.0) | 86 (5.3) | 85.7 (6.0) | 84.5 (6.5) | 91.8 (2.5)
  Week 3: Post-Dose (n= 10, 7, 7, 8, 10) | 90 (4.2) | 77.8 (4.3) | 75.7 (4.8) | 78.6 (6.4) | 80.7 (3.1)
  Week 4: Pre-Dose (n= 9, 7, 9, 9, 10) | 86.4 (3.6) | 81.8 (3.2) | 85.9 (5.2) | 81.2 (4.0) | 88.9 (3.0)
  Week 4: Post-Dose (n= 9, 6, 9, 8, 10) | 85.9 (3.4) | 75.1 (3.4) | 77.3 (5.0) | 71.6 (2.8) | 83.1 (3.8)
  Week 6: Pre-Dose (n= 9, 7, 8, 8, 8) | 87.9 (4.8) | 82.7 (3.7) | 81.6 (2.6) | 81.6 (4.7) | 91.3 (2.1)
  Week 6: Post-Dose (n= 9, 7, 8, 8, 8) | 85.4 (4.1) | 74.2 (3.4) | 74.4 (4.3) | 70.1 (3.4) | 83.3 (3.8)
  Week 8: Pre-Dose (n= 8, 6, 8, 8, 7) | 87.3 (5.3) | 85.2 (4.0) | 79.8 (3.2) | 83.7 (4.9) | 92 (4.4)
  Week 8: Post-Dose (n= 8, 6, 8, 8, 7) | 81.1 (5.0) | 78.7 (4.0) | 75.4 (4.4) | 75.3 (5.0) | 84.5 (5.2)
  Week 10: Pre-Dose (n= 8, 4, 7, 7, 6) | 88.7 (3.8) | 83.5 (2.2) | 86.2 (3.8) | 80.3 (5.1) | 93.4 (3.1)
  Week 10: Post-Dose (n= 8, 4, 7, 7, 6) | 83.2 (4.9) | 73.8 (1.5) | 81.3 (3.8) | 67 (3.7) | 84.2 (4.8)

7. Secondary Outcome: Change From Standing to Sitting Systolic Blood Pressure (SBP) at Week 10
Description: SBP is the BP (pressure exerted by circulating blood on the walls of blood vessels) when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle of heart. A total of 3 measurements were performed and average was calculated at each time point in participant's non-dominant arm using appropriate-sized cuff (cuff bladder encircling at least 80% of the arm). The same arm was used throughout the study.
Time Frame: Pre-Dose and 2 hours Post-Dose on Week 10
Population: FAS:all randomized participants who received study treatment at least twice after Placebo Run-in Phase, but not necessarily at 2 consecutive visits. "N" (number of participants analyzed): participants evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Number analyzed (Participants) | 7 | 4 | 7 | 7 | 6
mmHg
  Week 10: Pre-Dose | 1.32 (1.78) | 0.46 (2.34) | 1.67 (1.76) | -0.54 (1.74) | -0.85 (2.01)
  Week 10: Post-Dose | 2.63 (1.97) | -0.55 (2.59) | 1.28 (1.95) | -1.30 (1.93) | 1.66 (2.22)
Statistical Analysis 1: Comparison: Placebo vs TBC3711 10 mg; Pre-Dose on Week 10: p-value was obtained using an ANCOVA model on the sitting-standing difference at Week 10 (Pre-Dose) with the sitting-standing difference at Baseline as a covariate; Test type: Superiority or Other; p = 0.7758, ANCOVA; LS Mean Difference = 0.86, 95% CI 2-sided [-5.31 to 7.03], Standard Error of Mean 3.00
Statistical Analysis 2: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.8880, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-5.40 to 4.71], Standard Error of Mean 2.45
Statistical Analysis 3: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.4573, ANCOVA; LS Mean Difference = 1.86, 95% CI 2-sided [-3.21 to 6.93], Standard Error of Mean 2.46
Statistical Analysis 4: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.4424, ANCOVA; LS Mean Difference = 2.17, 95% CI 2-sided [-3.56 to 7.91], Standard Error of Mean 2.78
Statistical Analysis 5: Comparison: Placebo vs TBC3711 10 mg; Post-Dose on Week 10: p-value was obtained using an ANCOVA model on the sitting-standing difference at Week 10 (Post-Dose) with the sitting-standing difference at Baseline as a covariate; Test type: Superiority or Other; p = 0.3470, ANCOVA; LS Mean Difference = 3.18, 95% CI 2-sided [-3.65 to 10.01], Standard Error of Mean 3.32
Statistical Analysis 6: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.6249, ANCOVA; LS Mean Difference = 1.34, 95% CI 2-sided [-4.25 to 6.94], Standard Error of Mean 2.72
Statistical Analysis 7: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.1625, ANCOVA; LS Mean Difference = 3.92, 95% CI 2-sided [-1.69 to 9.54], Standard Error of Mean 2.73
Statistical Analysis 8: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.7556, ANCOVA; LS Mean Difference = 0.97, 95% CI 2-sided [-5.38 to 7.31], Standard Error of Mean 3.08

8. Secondary Outcome: Change From Standing to Sitting Diastolic Blood Pressure (DBP) at Week 10
Description: DBP is the BP (pressure exerted by circulating blood on the walls of blood vessels) when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles of heart. A total of 3 measurements were performed and average was calculated at each time point in participant's non-dominant arm using appropriate-sized cuff (cuff bladder encircling at least 80% of the arm). The same arm was used throughout the study.
Time Frame: Pre-Dose and 2 hours Post-Dose on Week 10
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Number analyzed (Participants) | 7 | 4 | 7 | 7 | 6
mmHg
  Week 10: Pre-Dose | -0.95 (0.95) | 2.04 (1.27) | -1.42 (0.95) | -1.18 (0.98) | -0.43 (1.03)
  Week 10: Post-Dose | -1.28 (1.32) | 1.50 (1.77) | -0.09 (1.32) | 0.68 (1.36) | 0.80 (1.43)
Statistical Analysis 1: Comparison: Placebo vs TBC3711 10 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0714, ANCOVA; LS Mean Difference = -2.99, 95% CI 2-sided [-6.25 to 0.28], Standard Error of Mean 1.59
Statistical Analysis 2: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.7269, ANCOVA; LS Mean Difference = 0.47, 95% CI 2-sided [-2.29 to 3.24], Standard Error of Mean 1.34
Statistical Analysis 3: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.8656, ANCOVA; LS Mean Difference = 0.23, 95% CI 2-sided [-2.58 to 3.04], Standard Error of Mean 1.36
Statistical Analysis 4: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.7113, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-3.41 to 2.36], Standard Error of Mean 1.40
Statistical Analysis 5: Comparison: Placebo vs TBC3711 10 mg; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.2204, ANCOVA; LS Mean Difference = -2.77, 95% CI 2-sided [-7.32 to 1.77], Standard Error of Mean 2.21
Statistical Analysis 6: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.5298, ANCOVA; LS Mean Difference = -1.19, 95% CI 2-sided [-5.04 to 2.66], Standard Error of Mean 1.87
Statistical Analysis 7: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.3135, ANCOVA; LS Mean Difference = -1.95, 95% CI 2-sided [-5.86 to 1.96], Standard Error of Mean 1.90
Statistical Analysis 8: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.2962, ANCOVA; LS Mean Difference = -2.08, 95% CI 2-sided [-6.09 to 1.93], Standard Error of Mean 1.95

9. Secondary Outcome: Change From Pre-Dose to Post-Dose in Systolic Blood Pressure (SBP) at Week 10
Description: as for outcome 7
Time Frame: Pre-Dose and 2 hours Post-Dose on Week 10
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Number analyzed (Participants) | 7 | 4 | 7 | 7 | 6
mmHg
  Week 10: Sitting | -8.33 (3.23) | -4.59 (4.30) | -4.49 (3.25) | -5.87 (3.23) | -7.03 (3.53)
  Week 10: Standing | -7.34 (2.95) | -4.41 (4.19) | -3.13 (3.16) | -5.24 (3.17) | -11.17 (3.42)
Statistical Analysis 1: Comparison: Placebo vs TBC3711 10 mg; Week 10 Sitting: p-value was obtained using an ANCOVA model on the post-dose minus pre-dose difference at Week 10 with the post-dose minus pre-dose difference at Baseline as a covariate; Test type: Superiority or Other; p = 0.4933, ANCOVA; LS Mean Difference = -3.74, 95% CI 2-sided [-14.84 to 7.35], Standard Error of Mean 5.39
Statistical Analysis 2: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.4080, ANCOVA; LS Mean Difference = -3.85, 95% CI 2-sided [-13.26 to 5.57], Standard Error of Mean 4.57
Statistical Analysis 3: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.5936, ANCOVA; LS Mean Difference = -2.47, 95% CI 2-sided [-11.86 to 6.93], Standard Error of Mean 4.56
Statistical Analysis 4: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.7883, ANCOVA; LS Mean Difference = -1.30, 95% CI 2-sided [-11.17 to 8.57], Standard Error of Mean 4.79
Statistical Analysis 5: Comparison: Placebo vs TBC3711 10 mg; Week 10 Standing: p-value was obtained using an ANCOVA model on the post-dose minus pre-dose difference at Week 10 with the post-dose minus pre-dose difference at Baseline as a covariate; Test type: Superiority or Other; p = 0.5719, ANCOVA; LS Mean Difference = -2.93, 95% CI 2-sided [-13.46 to 7.60], Standard Error of Mean 5.12
Statistical Analysis 6: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.3401, ANCOVA; LS Mean Difference = -4.21, 95% CI 2-sided [-13.11 to 4.70], Standard Error of Mean 4.33
Statistical Analysis 7: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.6329, ANCOVA; LS Mean Difference = -2.10, 95% CI 2-sided [-11.01 to 6.82], Standard Error of Mean 4.34
Statistical Analysis 8: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.4037, ANCOVA; LS Mean Difference = 3.83, 95% CI 2-sided [-5.45 to 13.11], Standard Error of Mean 4.51

10. Secondary Outcome: Change From Pre-Dose to Post-Dose in Diastolic Blood Pressure (DBP) at Week 10
Description: as for outcome 8
Time Frame: Pre-Dose and 2 hours Post-Dose on Week 10
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Number analyzed (Participants) | 7 | 4 | 7 | 7 | 6
mmHg
  Week 10: Sitting | -8.57 (2.50) | -9.79 (3.26) | -3.69 (2.46) | -11.28 (2.52) | -7.23 (2.66)
  Week 10: Standing | -6.90 (2.44) | -10.35 (3.36) | -5.51 (2.55) | -11.67 (2.61) | -7.97 (2.78)
Statistical Analysis 1: Comparison: Placebo vs TBC3711 10 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.7685, ANCOVA; LS Mean Difference = 1.21, 95% CI 2-sided [-7.19 to 9.62], Standard Error of Mean 4.08
Statistical Analysis 2: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.1739, ANCOVA; LS Mean Difference = -4.88, 95% CI 2-sided [-12.07 to 2.30], Standard Error of Mean 3.49
Statistical Analysis 3: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.4612, ANCOVA; LS Mean Difference = 2.71, 95% CI 2-sided [-4.74 to 10.15], Standard Error of Mean 3.61
Statistical Analysis 4: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.7172, ANCOVA; LS Mean Difference = -1.34, 95% CI 2-sided [-8.90 to 6.21], Standard Error of Mean 3.67
Statistical Analysis 5: Comparison: Placebo vs TBC3711 10 mg; [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.4098, ANCOVA; LS Mean Difference = 3.45, 95% CI 2-sided [-5.01 to 11.91], Standard Error of Mean 4.12
Statistical Analysis 6: Comparison: Placebo vs TBC3711 50 mg; [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.6943, ANCOVA; LS Mean Difference = -1.38, 95% CI 2-sided [-8.54 to 5.78], Standard Error of Mean 3.48
Statistical Analysis 7: Comparison: Placebo vs TBC3711 100 mg; [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.2042, ANCOVA; LS Mean Difference = 4.78, 95% CI 2-sided [-2.76 to 12.31], Standard Error of Mean 3.67
Statistical Analysis 8: Comparison: Placebo vs TBC3711 200 mg; [analysis description as in outcome 9, analysis 5]; Test type: Superiority or Other; p = 0.7791, ANCOVA; LS Mean Difference = 1.07, 95% CI 2-sided [-6.69 to 8.83], Standard Error of Mean 3.77

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | TBC3711 10 mg | TBC3711 50 mg | TBC3711 100 mg | TBC3711 200 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 1/11 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 3/8 | 3/11 | 4/10 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | TBC3711 10 mg (N=8) | TBC3711 50 mg (N=11) | TBC3711 100 mg (N=10) | TBC3711 200 mg (N=10)
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | TBC3711 10 mg (N=8) | TBC3711 50 mg (N=11) | TBC3711 100 mg (N=10) | TBC3711 200 mg (N=10)
Fatigue (General disorders) | 0 | 1 | 0 | 2 | 0
Oedema peripheral (General disorders) | 2 | 0 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 0 | 1 | 2
Dyspnoea (Nervous system disorders) | 0 | 0 | 2 | 0 | 1

LIMITATIONS AND CAVEATS:
Results for 'change from standing to sitting SBP and DBP' and 'change from pre-dose to post-dose SBP and DBP' are reported only at Week 10 as per changes in planned analysis because of early termination of the study and clinical development program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.